CLINICAL TRIAL: NCT03628157
Title: Ridge Augmentation in Atrophic Anterior Maxillary Ridges With a Titanium Reinforced Polytetraflouroethelene Membrane and Anorganic Bovine Bone-Derived Mineral With and Without Particulated Autogenous Bone Chips
Brief Title: GBR With Ptfe With Bovine Bone With and Without Autogenous
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif osama hegazy, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Bone augmentation
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Atrophied Anterior Maxillary Ridges

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- intervention (Experimental): using a bio-oss bovine bone alone
  Interventions: Other: Geistlich Bio-Oss® bovine bone alone
- control (Active Comparator): using a bio-oss bovine bone with autogenous bone ratio 1:1
  Interventions: Other: Geistlich Bio-Oss® bovine bone alone

INTERVENTIONS:
Other: Geistlich Bio-Oss® bovine bone alone — Ridge augmentation by titanium reinforced polytetraflouroethelene membrane and anorganic bovine bone derived mineral alone

SUMMARY:
Ridge Augmentation in Atrophic Anterior Maxillary Ridges with a Titanium Reinforced Polytetraflouroethelene Membrane and Anorganic Bovine Bone-Derived Mineral in intervention group and Anorganic Bovine Bone-Derived Mineralwith Particulated Autogenous Bone Chips in control group.

CBCT will be done before surgery, immediate after surgery and 6 month to compare the bone gain in mm.

Bone sample will be collected during exposure after 6 month of surgery by trephine bur to assess the bone quality through histo-morphometric analysis in order to determine the size, shape and orientation of the bony trabeculae, the size and porosity of the bony cortex in addition to the new bone/ bone substitute ratio

* 1ry outcome: Amount of bone gain will be measured using linear measurements from CBCT immediate after surgery and after 6 month.
* 2ry outcome: a bone sample will be collected and analyzed under histo-morphometric analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with atrophied anterior maxillary ridge area.

  * Age: 18 years and older.
  * Both sexes.
  * No intraoral soft and hard tissue pathology.
  * No systemic condition that contraindicate bone augmentation

Exclusion Criteria:

* • Heavy smokers more than 20 cigarettes per day.(32)

  * Patients with systemic disease that may affect normal healing.
  * Psychiatric problems.
  * Disorders to bone augmentation are related to history of radiation therapy to the head and neck neoplasia.
  * Pregnant or nursing women.
  * Patients with uncontrolled diabetes mellitus, rheumatoid arthritis or osteoporosis.
  * Patient with previous history of radiotherapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Amount of bone gain (height and width in mm) | 6 months
  will be measured using linear measurements from CBCT

SECONDARY OUTCOMES:
a bone sample will be collected and analyzed under histo-morphometric analysis. (no of bone cells in cubic mm) | 6 months
  a bone sample will be collected and analyzed under histo-morphometric analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No